CLINICAL TRIAL: NCT06223451
Title: Evaluation of the Efficacy of Low-Frequency Repetitive Transcranial Magnetic Stimulation on Unilateral Neglect in Patients With Subacute-Chronic Phase After Ischemic Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Ayşenur Mert, Medical doctor, Ankara City Hospital Bilkent
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10026592
Record Dates: First submitted 2024-01-04; First posted 2024-01-25 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Neglect, Hemispatial
Keywords: İskemic stroke; Transcranial magnetic stimulation; Unilateral neglect
MeSH Terms: conditions — Perceptual Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active repetitive transcranial magnetic stimulation in stroke patients with unilateral neglect. (Active Comparator): Inhibitory repetitive transcranial magnetic stimulation will be applied to 11 patients with unilateral neglect due to ischemic stroke under the supervision of a doctor for a total of 10 sessions over 2 weeks with conventional rehabilitation. Each session will last for 20 minutes,total of 1200 pulses, 1 Hz repetitive transcranial manyetic stimulation over the unaffected left posterior parietal cortex.
  Interventions: Device: Active Repetitive Transcranial Magnetic Stimulation
- Sham repetitive transcranial magnetic stimulation in stroke patients with unilateral neglect. (Sham Comparator): Patients in the sham group will receive sham transcranial magnetic stimulation with sham coil for 20 minutes a day, 10 sessions in total, together with conventional rehabilitation.
  Interventions: Device: Sham Repetitive Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Active Repetitive Transcranial Magnetic Stimulation — Repetitive Transcranial Magnetic Stimulation (rTMS) is a non-invasive brain stimulation method that can alter the excitability of the motor area by generating a magnetic field through a coil. Low-frequency stimulation (<1 Hz) applied with rTMS has inhibitory effects. Repetitive transcranial magnetic stimulation has a neurorehabilitative role as it can modulate the excitability of targeted brain areas. Inhibitory repetitive transcranial magnetic stimulation will be applied to 11 patients with unilateral neglect due to ischemic stroke under the supervision of a doctor for a total of 10 sessions over 2 weeks with conventional rehabilitation.Each session will last for 20 minutes,total of 1200 pulses, 1 Hz repetitive transcranial manyetic stimulation over the unaffected left posterior parietal cortex.
  Arms: Active repetitive transcranial magnetic stimulation in stroke patients with unilateral neglect.
Device: Sham Repetitive Transcranial Magnetic Stimulation — Patients in the sham group will receive sham transcranial magnetic stimulation with sham coil for 20 minutes a day, 10 sessions in total, together with conventional rehabilitation.
  Arms: Sham repetitive transcranial magnetic stimulation in stroke patients with unilateral neglect.

SUMMARY:
The aim of this study was to randomize stroke patients with unilateral neglect into 2 groups, active and sham groups, and to examine the effects of active inhibitory repetitive transcranial magnetic stimulation on the reduction of neglect symptoms, functional recovery and independence of these patients in activities of daily living.

DETAILED DESCRIPTION:
Patients diagnosed with ischemic stroke at least 1 month ago, with unilateral neglect, receiving inpatient rehabilitation at stroke clinics, and meeting the study criteria for both genders between the ages of 18-80, will be divided into two groups. A total of 22 stroke patients, informed about the applied treatments and potential risks, and providing written consent, will be randomly assigned to receive either active repetitive transcranial magnetic stimulation (rTMS) combined with conventional rehabilitation (Mirror therapy and Visual scanning training) or sham (imitation) repetitive transcranial magnetic stimulation (rTMS) combined with conventional rehabilitation.

The study will include 22 randomly selected patients with neglect, with 11 planned in the intervention group and 11 in the control group. Patients will receive active rTMS or sham rTMS for a total of 10 sessions, each lasting 20 minutes, alongside conventional rehabilitation over a period of 2 weeks. rTMS applications will be conducted once daily before the daily rehabilitation program.

ELIGIBILITY:
Inclusion Criteria:

* First-time ischemic stroke
* Patients at least 1 month after the stroke
* To be aged between 18 and 80 years old
* Presence of unilateral neglect
* No significant cognitive impairment (MMSE > 24 points)
* Signing an informed consent form indicating willingness to participate in the study

Exclusion Criteria:

* Epilepsy, history of seizure
* Metallic implant in the area of stimulation (cochlear implant, brain pacemaker, drug pump etc.)
* Presence of cardiac pacemaker
* Severe general condition disorder or accompanying neurological disease
* Aphasi
* Pregnancy
* Under 18 years of age and over 80 years of age
* Visual impairment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2023-06-15 (Actual); Primary Completion 2024-02-15 (Actual); Study Completion 2024-04-15 (Actual)

PRIMARY OUTCOMES:
Star Cancellation Test | Before treatment(initial), two weeks after the beginning of the treatment, four weeks after the beginning of the treatment, six weeks after the beginning of the treatment
  The star cancellation test, there are 13 letters and 10 short words placed between 52 large and 56 small stars. The patient is required to mark all the small stars using a pencil. To demonstrate how it should be done, two small stars are selected from the central section.Scores are calculated by identifying the ratio of the number of removed small stars/the total number of small stars 100 for each empty half-space on the left and right sides.
Line Bisection Test | Before treatment(initial), two weeks after the beginning of the treatment, four weeks after the beginning of the treatment, six weeks after the beginning of the treatment
  The Line Bisection Test is a rapid measure to detect the presence of unilateral spatial neglect. To complete the test, a pencil mark is placed in the middle of 18 horizontal lines. The test is scored by measuring the deviation from the actual center of the line.

SECONDARY OUTCOMES:
Catherine Bergego Scale | Before treatment(initial), two weeks after the beginning of the treatment, four weeks after the beginning of the treatment, six weeks after the beginning of the treatment
  Catherine Bergego Scale: Analyzes the functioning of the neglect patient in daily life situations. Each question is scored from zero to three, where 0 corresponds to the absence of neglect for the given task; 1 represents mild neglect, 2 represents moderate neglect, and 3 corresponds to severe unilateral neglect. If the total score is between 1 and 10, it is considered mild neglect; if it is between 11 and 20, it is considered moderate neglect; and if it is between 21 and 30, it is considered severe neglect.
Stroke Impact Scale | Before treatment(initial), two weeks after the beginning of the treatment, four weeks after the beginning of the treatment, six weeks after the beginning of the treatment
  This scale, which aims to assess the quality of life after stroke by patients themselves or their caregivers, consists of 8 subsections and 59 questions. Each question is scored by evaluating the difficulty experienced in the last week by giving 5 points. The total score ranges from 0-100 and a high score indicates improvement in stroke patients.
Mini-Mental State Examination | Before treatment(initial), two weeks after the beginning of the treatment, four weeks after the beginning of the treatment, six weeks after the beginning of the treatment
  It is a screening test used to assess the cognitive status of patients. It is categorized under 5 main headings: orientation, recording memory, attention and calculation, recall and language. It is evaluated over a total of 30 points.
Brunnstrom Recovery Stage | Before treatment(initial), two weeks after the beginning of the treatment, four weeks after the beginning of the treatment, six weeks after the beginning of the treatment
  The test is used to assess post-stroke motor recovery. The motor development stages of hemiplegic patients are graded on a scale of 1-6.stage 1 flaccid period is rated as the worst stage, stage 6 is rated as the best stage with isolated movements.

CONTACTS AND LOCATIONS:
Overall Officials: Ayşenur Mert Kurt, Medical Doctor, Principal Investigator — Ankara City Hospital Bilkent; Zeynep A Kurtaran, Professor Doctor, Study Director — Ankara City Hospital Bilkent
Locations (1):
- Ankara Bilkent City Hospital Physical Therapy and Rehabilitation Hospital, Ankara, Bilkent-Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cha HG, Kim MK. The effects of repetitive transcranial magnetic stimulation on unilateral neglect of acute stroke patients: A randomised controlled trial. Hong Kong Physiother J. 2015 Dec;33(2):53-58. doi: 10.1016/j.hkpj.2015.04.001. Epub 2015 Jun 12. PMID 30930568
- [Result] Brighina F, Bisiach E, Oliveri M, Piazza A, La Bua V, Daniele O, Fierro B. 1 Hz repetitive transcranial magnetic stimulation of the unaffected hemisphere ameliorates contralesional visuospatial neglect in humans. Neurosci Lett. 2003 Jan 16;336(2):131-3. doi: 10.1016/s0304-3940(02)01283-1. PMID 12499057
- [Result] Kim YK, Jung JH, Shin SH. A comparison of the effects of repetitive transcranial magnetic stimulation (rTMS) by number of stimulation sessions on hemispatial neglect in chronic stroke patients. Exp Brain Res. 2015 Jan;233(1):283-9. doi: 10.1007/s00221-014-4112-9. Epub 2014 Oct 21. PMID 25332169